CLINICAL TRIAL: NCT01422330
Title: An Open-Label Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Etravirine (ETR) in Combination With Other Antiretrovirals (ARVs) in Antiretroviral Treatment-Experienced HIV-1 Infected Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Etravirine Administered in Combination With Other Antiretroviral Agents in Antiretroviral Treatment-Experienced HIV-1 Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017860; TMC125IFD3002 (Other: Janssen R&D Ireland); 2010-023532-16 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2011-08-23 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
Keywords: Human Immunodeficiency Virus (HIV) infection; TMC125IFD3002; TMC125; Intelence; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etravirine (Experimental)
  Interventions: Drug: Etravirine

INTERVENTIONS:
Drug: Etravirine — Type=exact number, unit=mg, number=100, form=tablet, route=oral use, 2 tablets. Type=exact number, unit=mg, number=200, form=tablet, route=oral use, 1 tablet. The drug is taken twice a day, after meals.

SUMMARY:
The purpose of this study is to learn more about the safety and tolerability of etravirine. Etravirine is a type of non-nucleoside reverse transcriptase inhibitor (NNRTI) which has shown high activity against wild-type human immunodeficiency virus (HIV-1), and HIV strains resistant to other non-nucleotide agents.

DETAILED DESCRIPTION:
This is an open-label (all people involved know the identity of the intervention), single arm, multicenter Phase IV study to evaluate the safety, tolerability, and pharmacokinetics of etravirine (ETR) in combination with antiretroviral (ARV) therapy other than darunavir (DRV) + ritonavir (rtv). In addition, the antiviral activity and the pharmacokinetic/pharmacodynamic profile, and safety of ETR will be assessed. The study will consist of a screening period of maximum 6 weeks, a baseline visit, and a 48-week treatment period. After the end of the treatment period, patients with ongoing adverse events (AEs) will be followed for an additional 4 weeks. At least 200 ARV treatment-experienced human immunodeficiency virus (HIV-1) infected patients will be enrolled in this study. Patients will be considered ARV treatment-experienced if they have been on their current stable highly active antiretroviral therapy (HAART) regimen for at least 8 weeks prior to screening. The study population will consist of patients who need to change their current HAART regimen due to any of the following reasons: (1) patients experiencing virologic failure (with a screening viral load value >=500 HIV-1 RNA copies/mL), or (2) patients switching due to simplification of their current regimen or due to AEs and/or tolerability reasons (with a screening viral load value <50 HIV-1 RNA copies/mL). Patients will receive ETR 200 mg twice daily in combination with an investigator-selected background regimen. In addition to ETR, which needs to be active based on resistance testing, the background regimen should consist of at least 1 active ARV resulting in a treatment regimen with at least 2 active ARVs. The following exceptions to this are: (1) if raltegravir (RAL) or atazanavir/ritonavir (ATV/rtv) are part of the background regimen, the number of active ARVs in this background regimen should be at least 2; (2) low-dose ritonavir should not be counted as an active ARV. DRV/rtv will not be allowed in the background regimen in order to evaluate the safety and pharmacokinetics of ETR in combination with ARVs other than DRV/rtv. Furthermore, a background regimen consisting of nucleoside transcriptase inhibitors (NRTIs) only will not be allowed. The background regimen cannot be modified until the end of the treatment period with the following exception: switches within the ARV class will be allowed for well documented tolerability/toxicity reasons. For patients who, in the opinion of the investigator, are deriving clinical benefit from ETR, and to whom ETR is not commercially available in his/her country, is not reimbursed or cannot be accessed from another source (e.g., access program, government program) in the region the patient is living in, the possibility to extend their ETR treatment period will be provided. The ETR tablets are to be taken orally twice daily after a meal. A total daily dose of 400 mg is to be taken for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Treatment with current stable HAART for at least 8 weeks prior to screening
* Currently experiencing virologic failure (screening viral load value >=500 HIV-1 RNA copies /mL), or switching due to simplification of their regimen or due to adverse event or tolerability reasons, (screening viral load value <50 HIV-1 RNA copies /mL)
* Demonstrated sensitivity to etravirine and to at least 1 antiretroviral (ARV) agent in the background regimen, based on the resistance test at screening or resistance history or have previously received treatment with etravirine
* Patients agree not to have unprotected sex while on the study
* No currently active AIDS-defining illness
* Did not take any non-ARV investigational agents within 90 days prior to screening
* No use of disallowed treatments
* Adequate liver function

Exclusion Criteria:

* Any currently active illness or toxicity due to HIV infection
* Any active clinically significant disease or findings during screening of medical history or physical examination that, in the investigator's opinion, would compromise the patient's safety or outcome of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with an Adverse Event (AEs) | 48 weeks

SECONDARY OUTCOMES:
Proportion of Participants with Virologic Suppression [Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) less than (<) 50 copies/Milliliter (mL)] at Week 48 | 48 weeks
  Food and Drug Administration (FDA) Snapshot analysis is based on the last observed viral load (VL) data within the Week 48 window: virologic response is defined as HIV-1 RNA<50 copies/mL (observed case); missing HIV-1 RNA is considered as non-response.
Changes in CD4 Cell Count at Week 48 | 48 weeks
Changes in Viral Genotype/Phenotype Over Time | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (42):
- United States (9):
  - Phoenix, Arizona
  - Beverly Hills, California
  - North Hollywood, California
  - Fort Laudersale, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Springfield, Massachusetts
  - Akron, Ohio
  - Longview, Texas
- Argentina (2):
  - Buenos Aires
  - Rosario
- France (2):
  - Le Kremlin-Bicêtre
  - Paris
- Guatemala City, Guatemala
- Mexico (2):
  - Guadalajara
  - México
- Peru (2):
  - Iquitos
  - Lima
- San Juan, Puerto Rico
- Romania (4):
  - Brasov
  - Constanța
  - Craiova
  - Timișoara
- Russia (6):
  - Krasnodar
  - Moscow
  - Saint Petersburg
  - Smolensk
  - Volgograd
  - Voronezh
- South Africa (9):
  - Bloemfontein
  - Boksburg
  - Dundee
  - Durban
  - Johannesburg
  - Newtown
  - Port Elizabeth
  - Pretoria
  - Westdene Johannesburg Gauteng
- Ukraine (4):
  - Donetsk
  - Kyiv
  - Luhansk
  - Sumy

REFERENCES:
- [Derived] Arathoon E, Bhorat A, Silaghi R, Crauwels H, Lavreys L, Tambuyzer L, Vanveggel S, Opsomer M. Week 48 results of a Phase IV trial of etravirine with antiretrovirals other than darunavir/ritonavir in HIV-1-infected treatment-experienced adults. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19783. doi: 10.7448/IAS.17.4.19783. eCollection 2014. PMID 25397527
- See also: An Open-Label Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Etravirine (ETR) in Combination With Other Antiretrovirals (ARVs) in Antiretroviral Treatment-Experienced HIV-1 Infected Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1100&filename=CR017860_CSR.pdf